CLINICAL TRIAL: NCT01775631
Title: A Phase 1b, Open-label, Multicenter Study of Urelumab (BMS-663513) in Combination With Rituximab in Subjects With Relapsed/Refractory B-cell Malignancies
Brief Title: Combination Study of Urelumab and Rituximab in Patients With B-cell Non-Hodgkins Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA186-017
Record Dates: First submitted 2013-01-23; First posted 2013-01-25 (Estimated); Last update posted 2017-03-31 (Actual); Status verified 2016-09

CONDITIONS: B-Cell Malignancies
MeSH Terms: interventions — urelumab; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm -1 - Urelumab + Rituximab (Experimental): Urelumab (BMS-663513) flat dose intravenous infusion on specified days
  Rituximab intravenous flat dose infusion on specified days
  Interventions: Biological: Urelumab; Biological: Rituximab
- Arm 1 - Urelumab + Rituximab (Experimental): Urelumab (BMS-663513) flat dose intravenous infusion on specified days
  Rituximab intravenous flat dose infusion on specified days
  Interventions: Biological: Urelumab; Biological: Rituximab

INTERVENTIONS:
Biological: Urelumab
  Other Names: BMS-663513
Biological: Rituximab

SUMMARY:
The purpose of the study is to determine the safety, tolerability and maximum tolerated dose of Urelumab in combination with Rituximab in patients with B-cell Non-Hodgkins Lymphoma

DETAILED DESCRIPTION:
Intervention model: Dose Escalation (part 1) of study= Sequential Design; Dose Expansion (part 2) of study= Parallel Design

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com.

Inclusion Criteria:

* Clinical diagnosis of relapsed/refractory B-cell Malignancies (B-Non-Hodgkins Lymphoma (NHL)) per International Workshop Group (IWG)
* Progressed or refractory to at least 1 prior line of standard therapy
* Subjects in Expansion cohorts are restricted to relapsed/refractory diffuse large B-cell lymphoma (DLBCL) or Follicular Lymphoma (FL) subjects who are either relapsed or refractory to prior rituximab or ritxumab-containing chemotherapy regimens
* Follicular Lymphoma (FL) must have at least 1 lesion that can be biopsied at screening and on treatment
* Eastern Cooperative Oncology Group (ECOG) of 0 to 1

Exclusion Criteria:

* Active or progressing brain metastases
* Other concomitant malignancies (with some exceptions per protocol)
* Active or history of autoimmune disease
* Positive test for human immunodeficiency virus (HIV) 1&2 or known Acquired immune deficiency syndrome (AIDS)
* History of any hepatitis (A, B or C)
* History of grade 3-4 drug-related hepatitis
* Known current drug or alcohol abuse
* Active tuberculosis (TB)
* Prior therapy with any antibody/drug that targets the T cell coregulatory proteins, including but not limited to, anti-CD137, Anti Cytotoxic T lymphocyte-associated antigen 4 (anti-CTLA4) or Anti-Glucocorticoid-induced tumor necrosis factor receptor (anti-GITR). However, Anti-Programmed Death-1 (anti-PD-1), Anti-Programmed Death-Ligand1 (anti-PD-L1) are permissible as prior therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2013-03; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of Urelumab in combination with Rituximab as measured by incidence of adverse events (AEs), serious AEs, death, vital sign changes, electrocardiograms (ECGs), physical examination results, and laboratory test abnormalities | Up to 60 days after last dose of Urelumab
Safety and tolerability of Urelumab in combination with Rituximab as measured by incidence of adverse events (AEs), serious AEs, death, vital sign changes, electrocardiograms (ECGs), physical examination results, and laboratory test abnormalities | Up to 110 days after last dose of Rituximab

SECONDARY OUTCOMES:
Efficacy-Antitumor Activity of Urelumab in combination with Rituximab as measured by best overall response, progression-free survival, time to response, and duration of response | Up to approximately 3 years
Maximum observed serum concentration (Cmax) of Urelumab and Rituximab | 12 time points up to Day 60 of Follow-up
Time of maximum observed serum concentration (Tmax) of Urelumab | 12 time points up to Day 60 of Follow-up
Area under the serum concentration-time curve from time zero to time of last quantifiable concentration (AUC(0-T)) of Urelumab | 12 time points up to Day 60 of Follow-up
Trough observed serum concentration (Cmin) of Urelumab and Rituximab | 12 + 9 time points up to Day 60 of Follow-up
Area under the concentration-time curve (AUC) in one dosing interval (AUC(TAU)) of Urelumab | 12 time points up to Day 60 of Follow-up
Immunogenicity of Urelumab in combination with Rituximab as determined by blood sample measurements of anti-drug antibodies (ADA) | Up to approximately 110 days post study drug

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (15):
- United States (15):
  - Ucla Department Of Medicine, Los Angeles, California
  - Stanford University Medical Center, Stanford, California
  - University Of Miami Sylvester Comprehensive Cancer Center, Miami, Florida
  - Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - University Of Iowa Hospitals And Clinics, Iowa City, Iowa
  - Dana Faber Cancer Institute, Boston, Massachusetts
  - University Of Michigan Health System, Ann Arbor, Michigan
  - Karmanos Cancer Institute, Detroit, Michigan
  - John Theurer Cancer Center, Hackensack, New Jersey
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - Providence Cancer Center Oncology And Hematology Care- Eastside, Portland, Oregon
  - Hospital Of The University Of Pennsylvania, Philadelphia, Pennsylvania
  - The University Of Texas Md Anderson Cancer Center, Houston, Texas
  - University Of Virginia School Of Medicine, Charlottesville, Virginia

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx